CLINICAL TRIAL: NCT01411865
Title: Evaluation of a Toolkit to Improve Cardiovascular Disease Screening and Treatment for People With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Shah-2
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus; Cardiovascular Disease
Keywords: Pragmatic randomized controlled trial; Cardiovascular risk reduction; Knowledge translation; Clinical practice guidelines; Administrative databases
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Toolkit
- Control (Other)
  Interventions: Other: Control

INTERVENTIONS:
Other: Toolkit — Cardiovascular Disease Toolkit mailed by the Canadian Diabetes Association to family physicians, accompanying the Spring/Summer 2009 edition of the quarterly newsletter, Canadian Diabetes. (Mailed in June 2009.) The Toolkit includes a summary of selected sections of the practice guidelines targeted towards primary care physicians; a synopsis of the key messages pertaining to cardiovascular disease risk; a laminated card with a simplified algorithm for cardiovascular risk assessment and treatment; and a pad of tear-off sheets for patients with a cardiovascular risk self-assessment tool.
  Arms: Intervention
Other: Control — The Spring/Summer 2009 issue of the quarterly newsletter, Canadian Diabetes, mailed on its own. The Cardiovascular Toolkit was mailed with the May 2010 issue of the newsletter.
  Arms: Control

SUMMARY:
Diabetes is a common and serious chronic disease. However, there is a large gap between the level of care that people should receive (based on research and guidelines) and the level of care they actually receive. With the release of their 2008 Clinical Practice Guidelines, the Canadian Diabetes Association has a strategy to improve heart disease screening and treatment for people with diabetes. This study will evaluate whether the strategy works. The focus of the strategy was to give all family physicians in Canada a Toolkit in June 2009 to help them delivery better care for their diabetic patients. In Ontario, only half of doctors received this Toolkit. We will compare the quality of care received by diabetic patients whose doctors received this Toolkit versus those who doctors did not.

DETAILED DESCRIPTION:
A cardiovascular disease Toolkit was developed by the Canadian Diabetes Association and mailed to family physician with the Spring/Summer 2009 edition of the newsletter, Canadian Diabetes. The Toolkit was packaged in a brightly-coloured box with Canadian Diabetes Association branding, and contained: 1) an introductory letter from the Chair of the practice guidelines' Dissemination and Implementation Committee; 2) an eight page summary of selected sections of the practice guidelines targeted towards primary care physicians; 3) a four page synopsis of the key guideline elements pertaining to cardiovascular disease risk; 4) a small double-sided laminated card with a simplified algorithm for cardiovascular risk assessment, vascular protection strategies and screening for cardiovascular disease; and 5) a pad of tear-off sheets for patients with a cardiovascular risk self-assessment tool and a list of recommended risk reduction strategies.

ELIGIBILITY:
Inclusion Criteria:

* Alive on 1 July 2009 with prevalent diabetes

Exclusion Criteria:

* Age <= 39
* Residing in long-term care

Secondary Analysis:

* Analysis will be repeated using all people alive on 1 July 2009 without prevalent diabetes using the same exclusion criteria, to determine the spill-over effect of the Intervention on physicians' other patients.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933789 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Death or non-fatal myocardial infarction | Up to 10 months

SECONDARY OUTCOMES:
Death, non-fatal myocardial infarction or non-fatal stroke | Up to 10 months
Death, non-fatal myocardial infarction, non-fatal stroke, or hospitalization for unstable angina or transient ischemic attack | Up to 10 months
Death | Up to 10 months
Hospitalization for myocardial infarction | Up to 10 months
Hospitalization for myocardial infarction or unstable angina | Up to 10 months
Hospitalization for stroke | Up to 10 months
Hospitalization for stroke or transient ischemic attack | Up to 10 months
Electrocardiogram | Up to 10 months
Cardiac stress test or nuclear imaging | Up to 10 months
Coronary angiography | Up to 10 months
Coronary revascularization procedure | Up to 10 months
Ambulatory cardiology or internal medicine visit | Up to 10 months
Prescription for angiotensin converting enzyme inhibitor or angiotensin receptor blocker | Up to 10 months
Prescription for at least one class of antihypertensive agent | Up to 10 months
Prescription for at least two classes of antihypertensive agents | Up to 10 months
Prescription for at least three classes of antihypertensive agents | Up to 10 months
Prescription for statin | Up to 10 months
Prescription for any glucose-lowering drug | Up to 10 months
Prescription for insulin | Up to 10 months
Prescription for nitrate | Up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Baiju R Shah, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Institute for Clinical Evaluative Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Result] Shah BR, Bhattacharyya O, Yu CH, Mamdani MM, Parsons JA, Straus SE, Zwarenstein M. Effect of an educational toolkit on quality of care: a pragmatic cluster randomized trial. PLoS Med. 2014 Feb 4;11(2):e1001588. doi: 10.1371/journal.pmed.1001588. eCollection 2014 Feb. PMID 24505216
- See also: Related study — http://clinicaltrials.gov/show/NCT01026688